CLINICAL TRIAL: NCT03359122
Title: Association of COPD Maintenance Medication Adherence With Resource Use and Cost Among COPD Patients-Retrospective Observational Cohort Study
Brief Title: Association of COPD Maintenance Medication Adherence With Resource Use and Cost Among COPD Patients
Acronym: MARU
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00123
Record Dates: First submitted 2017-11-08; First posted 2017-12-02 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the association of COPD maintenance inhalation medication (Inhaled Corticosteroid or ICS) adherence with COPD exacerbation healthcare resource utilization among COPD patients with exacerbation history.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to examine the association of COPD maintenance inhalation medication (Inhaled Corticosteroid or ICS) adherence with COPD exacerbation healthcare resource utilization among COPD patients with exacerbation history.

Study design: This study is a retrospective database analysis using 2014-2016 Guangzhou City health insurance database.

Data Source(s): Guangzhou city health insurance database will be used for this study. All outpatient and inpatient visits for one patient during 2014-2016 were available.

Study Population: This study will include patients with a physician COPD diagnosis in Guangzhou city health insurance database during 2015 and with complete treatment data during 1 year before and 1 year after the index date. The rough sample size of the study population was 49,000.

Outcome(s):

1. Indicators of COPD control: exacerbations;
2. Health resource utilization: annual number of inpatient days, inpatient visit number, emergency department (ED) visit number;
3. Costs: COPD exacerbation hospitalization expenditures, all-cause hospitalization expenditure.

Statistical Analysis:

Descriptive statistics will be used for all variables, as appropriate. Continuous variables will be summarized by the number of observations, mean, standard deviation, median, minimum, maximum, first quartile and third quartile. Categorical variables will be summarized by frequency counts and percentages at each category. Number of patients and number of missing for each variable will be summarized.

Logistic regression will be used to estimate the risk of any hospitalization. Generalized Linear Models (GLMs) with a gamma distribution and log link will be used to approximate the highly right-skewed distribution of medical expenditure.

For exploratory objectives, Propensity Score Matching (PSM) will be used to explore the association of medication class and health resource utilization if applicable. The interaction of medication class * adherence or subgroup analysis (by medication class) will be considered when conducting the regression model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COPD in 2015;
2. Patients had complete hospital visit data available during pre-index 1 year period and post 1 year follow-up;
3. Patients had at least one COPD exacerbation during 1 year prior to the index date;
4. Patients had at least 2 COPD maintenance medication claims during post index 1 year period, as 2 claims are recommended to calculate adherence.

Exclusion Criteria:

1. Inability to determine diagnoses from claims;
2. Individuals with other chronic respiratory conditions such as respiratory cancer, pulmonary fibrosis, asthma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients diagnosed with COPD in 2015 (a sub-group with exacerbation history will be used for primary, secondary and the first exploratory objectives analysis) and having continuous usage of COPD maintenance therapy during the 1 year follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 10067 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Indicators of COPD control | 2015.01-2016.12
  Number of exacerbations
Health resource utilization | 2015.01-2016.12
  Annual number of inpatient days
Costs of inpatient treatment | 2015.01-2016.12
  Cost of COPD exacerbation inpatient treatment
Health resource utilization | 2015.01-2016.12
  Inpatient visit number
Health resource utilization | 2015.01-2016.12
  Emergency department (ED) visit number
Costs of inpatient treatment | 2015.01-2016.12
  Cost of all-cause inpatient treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Beijing, China

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00123&attachmentIdentifier=763bcca5-a8d8-4c09-a11f-c96d64b435af&fileName=D2287R00123_Study_Report_Synopsis_MARU_26Jul2019.pdf&versionIdentifier=